CLINICAL TRIAL: NCT02775201
Title: A Comparison of Intra-operative and Ultrasound Guided Plantaris Release for the Treatment of Non-insertional Achilles Tendinopathy
Brief Title: Plantaris Release for Non-insertional Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fortius Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/0188
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Tendinopathy; Achilles Tendon
Keywords: plantaris; Tendinopathy; Achilles; Release
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plantaris release under ultrasound guidance (Active Comparator): Patients diagnosed with non-insertional Achilles tendinopathy will have plantaris released under ultrasound guidance by a consultant radiologist
  Interventions: Procedure: Plantaris excision surgically
- Plantaris excision surgically (Active Comparator): Patients diagnosed with non-insertional Achilles tendinopathy will have plantaris excised in surgery by a consultant orthopaedic surgeon
  Interventions: Procedure: Plantaris release under ultrasound guidance

INTERVENTIONS:
Procedure: Plantaris release under ultrasound guidance — In patients diagnosed with Achilles tendinopathy the plantaris tendon will be released using a small incision at the medial ankle under ultrasound guidance by a consultant radiologist
  Arms: Plantaris excision surgically
Procedure: Plantaris excision surgically — In patients diagnosed with Achilles tendinopathy the plantaris tendon will be excised in theatre by a consultant orthopaedic surgeon
  Arms: Plantaris release under ultrasound guidance

SUMMARY:
The plantaris tendon is recognised as an important factor in non-insertional Achilles tendinopathy (NIAT). A biomechanical study found the plantaris tendon is stiffer and stronger than the Achilles tendon (AT), thus reducing its capacity to elongate in response to loading. This is hypothesized to result in friction between the AT and plantaris in some NIAT patients. Current treatment is conservative management: physiotherapy and high volume injection of the paratenon. However 29% of patients fail to respond to conservative management and those with plantaris related symptoms require its surgical excision and stripping of the ventral aspect of the AT through a 3cm medial incision. This is performed in theatres under general anaesthetic with good or excellent results reported in 90% of cases.

Purely cutting the plantaris tendon using a minimally invasive endoscopic technique has also been successful. The plantaris tendon is easily visualized under ultrasound scan (USS) and tenotomy of tendons under USS guidance is performed elsewhere. Tenotomy of the plantaris tendon under USS guidance would necessitate a 5mm incision and may be performed under local anaesthetic as an out-patient. The current study thus plans a randomised clinical trial to compare outcomes (VISA-A scores and ultrasound tissue characterisation scans) from patients with NIAT undergoing plantaris release using an open surgical procedure with those undergoing a minimally invasive US guided procedure. The former is known to provide good clinical outcomes; however the latter could significantly reduce post-operative scarring, recovery times and costs. Findings will ensure ethical, quality and cost effective patient care.

DETAILED DESCRIPTION:
Midportion Achilles tendinopathy has been found to have an incidence of 1.85 per 1000 in the general population and is reported to be a career-ending condition in up to 5% of professional athletes. The mainstay of treatment at present is typically prescription of eccentric strengthening exercises, activity modification and analgesia. If conservative intervention fails then surgery can be indicated, and a wide range of different procedures are described. Open Achilles surgery may be successful in 75-100% of patients but debridement with excision of areas of tendinosis weakens the tendon and can delay return to sport for up to 18 months.

There is currently a growing acceptance for the role of the plantaris tendon in the development of medial Achilles tendon (AT) pain and focal medial Achilles tendinopathy. The plantaris arises from the lateral aspect of the supracondylar line of the femur, passing from lateral to medial deep to medial gastrocnemius and superficial to soleus, inserting into the medial aspect of the calcaneus. However there is wide variation in the exact insertion of the plantaris tendon observed distally. A large study examining 750 limbs reported 4 types of distal insertion, a further study reported 3 different insertion sites, whilst a more recent study reported 9 variations. Consistently 10-20% of plantaris tendons are identified to have a direct structural attachment to the AT. This variety of insertion patterns may explain why some individuals are more prone to plantaris issues than others.

Friction of the plantaris tendon against the medial border of the Achilles tendon and subsequent pain and swelling is a significant problem in elite track and field athletes, with an annual injury incidence of 3.9-9.3% reported. Biomechanical studies have hypothesized that this is due to the plantaris tendon being stiffer and stronger than the Achilles tendon (AT), thus reducing its capacity to elongate in response to loading. This is thought to cause friction between the AT and plantaris contributing to peritendon inflammation, which can induce tendinopathy changes to the AT through either a neuro-inflammatory mediation or via a compressive mechanism.

Twenty nine percent of patients with NIAT fail to respond to conservative management and many have to give up sporting activities. Patients who continue to experience symptoms may be referred for a high volume injection of the paratenon under ultrasound scan (USS) guidance - this aims to strip the paratenon layer from the AT which often becomes adherent with fibrous bands. This also strips the neovascularization from the ventral surface of the AT - this abnormal tissue has nerve fibres within it and it is believed that this is a major pain generator in NIAT. However, it is recognised that a sub-group of patients with NIAT have isolated medially-located pain approximately 4-6cm from insertion into the os calcis. On USS and Magnetic Resonance Imaging (MRI) the plantaris tendon may be seen to attach to the medial aspect of the AT (either inserting into the side of the AT directly rather than the os calcis or becoming adherent with fibrous tissue to the AT medial border). This is at the level of the AT where it has undergone a 90 degree rotation and corresponds to the soleus part of the tendon. Since the plantaris tendon crosses 2 joints (originating above the knee and inserting into the os calcis) whereas the soleus only crosses one joint (the ankle) there may be a differential movement of the plantaris against the medial border of the AT creating a frictional syndrome with subsequent focal inflammation and then tendinosis of the AT.

The treatment for this "plantaris syndrome" if it fails to respond to conservative measures or USS guided injections is to remove the plantaris tendon and surgically strip the ventral aspect of the AT through a 3cm medial incision. This is performed in theatres under general anaesthetic with good or excellent results being reported in 90% and 94% of professional athletes returning to sport.3 However, there have been papers reporting on the successful treatment of patients purely cutting the plantaris tendon using a minimally invasive endoscopic technique.The plantaris tendon is easily visualized under USS and tenotomy of tendons under USS guidance is described elsewhere. Performing a tenotomy of the plantaris tendon under USS guidance would necessitate a 5mm incision and may be performed under local anaesthetic as an out-patient. Currently it is not known whether this is as good as the open surgical procedure performed in theatre and the investigators would propose a randomized study comparing the techniques.

The rationale for the current study therefore is to compare clinical outcomes and AT structural changes in patients with NIAT undergoing plantaris excision using an open surgical procedure to those undergoing a minimally invasive US guided procedure performed in an out-patient clinic. The former is known to provide good clinical outcomes however the latter could significantly reduce post-operative scarring, recovery times and surgical costs. Thus, if found to be comparable, treating these patients in the clinic with an ultrasound guided plantaris release would offer a desirable alternative to surgery and result in a change of current clinical interventions for this population.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of medially located NIAT confirmed by USS and MRI.
2. Participants having undergone at least one course of conservative intervention including physiotherapy which has been unsuccessful.

Exclusion Criteria:

1. Any other co-existing lower limb injuries which would affect the outcome of patient reported outcome scores.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
VISA-A Questionnaire | 2 years
Ultrasound Tissue Characterisation | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fortius Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Andersson G, Danielson P, Alfredson H, Forsgren S. Nerve-related characteristics of ventral paratendinous tissue in chronic Achilles tendinosis. Knee Surg Sports Traumatol Arthrosc. 2007 Oct;15(10):1272-9. doi: 10.1007/s00167-007-0364-2. Epub 2007 Jun 29. PMID 17604979
- [Result] Calder JD, Freeman R, Pollock N. Plantaris excision in the treatment of non-insertional Achilles tendinopathy in elite athletes. Br J Sports Med. 2015 Dec;49(23):1532-4. doi: 10.1136/bjsports-2014-093827. Epub 2014 Nov 13. PMID 25394422
- [Result] Maffulli N, Spiezia F, Longo UG, Denaro V, Maffulli GD. High volume image guided injections for the management of chronic tendinopathy of the main body of the Achilles tendon. Phys Ther Sport. 2013 Aug;14(3):163-7. doi: 10.1016/j.ptsp.2012.07.002. Epub 2012 Nov 4. PMID 23131435
- [Result] Helms CA, Fritz RC, Garvin GJ. Plantaris muscle injury: evaluation with MR imaging. Radiology. 1995 Apr;195(1):201-3. doi: 10.1148/radiology.195.1.7892469.